CLINICAL TRIAL: NCT05846594
Title: An International Prospective Study to Evaluate the Impact of Liquid Biopsy in Participants With a Clinical Diagnosis of Advanced Cancer (L1ST)
Brief Title: A Study to Evaluate the Impact of Liquid Biopsy in Participants With a Clinical Diagnosis of Advanced Cancer
Acronym: L1st
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MO43989
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Lung Cancer; Metastatic Gastrointestinal Cancer
MeSH Terms: conditions — Lung Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Basic Workup: Metastatic Lung Cancer Cohort (Other): This cohort will enroll approximately 160 participants who have clinical evidence of de novo metastatic lung cancer and who have not had tissue biopsy performed prior to enrollment (classified as 'basic workup').
  Interventions: Diagnostic Test: FoundationOne® Liquid CDx Assay; Diagnostic Test: Standard of Care Diagnostic Pathway
- Basic Workup: Metastatic Gastrointestinal Cancer Cohort (Other): This cohort will enroll approximately 160 participants who have clinical evidence of de novo metastatic gastrointestinal cancer and who have not had tissue biopsy performed prior to enrollment (classified as 'basic workup').
  Interventions: Diagnostic Test: FoundationOne® Liquid CDx Assay; Diagnostic Test: Standard of Care Diagnostic Pathway
- Extended Workup: Metastatic Lung Cancer Cohort (Other): This cohort will enroll approximately 100 participants who have clinical evidence of de novo metastatic lung cancer and who have had tissue biopsy performed prior to enrollment (classified as 'extended workup').
  Interventions: Diagnostic Test: FoundationOne® Liquid CDx Assay; Diagnostic Test: Standard of Care Diagnostic Pathway
- Extended Workup: Metastatic Gastrointestinal Cancer Cohort (Other): This cohort will enroll approximately 100 participants who have clinical evidence of de novo metastatic gastrointestinal cancer and who have had tissue biopsy performed prior to enrollment (classified as 'extended workup').
  Interventions: Diagnostic Test: FoundationOne® Liquid CDx Assay; Diagnostic Test: Standard of Care Diagnostic Pathway

INTERVENTIONS:
Diagnostic Test: FoundationOne® Liquid CDx Assay — Participants will undergo liquid biopsy (FoundationOne® Liquid CDx) on blood samples collected once they have a clinical diagnosis of advanced cancer (as per label). Blood samples will be tested using the FoundationOne® Liquid CDx assay at a central laboratory. Results of the FoundationOne® Liquid CDx assay will be provided to the investigator to be used in accordance with professional guidelines in oncology for patients with malignant neoplasms.
Diagnostic Test: Standard of Care Diagnostic Pathway — Participants will undergo the local standard of care diagnostic pathway including tissue biopsy/standard of care (if tissue not available), pathology workup, and molecular workup, according to ESMO guidelines or national guidelines for each tumor type included in this study.

SUMMARY:
This is an international, prospective study to assess the impact of concomitant early use of liquid biopsy (FoundationOne® Liquid CDx) within the diagnostic pathway, compared with the standard of care diagnostic pathway, on the timing of routine cancer care in treatment-naïve participants presenting with a clinical diagnosis of advanced cancer, where the pathologic diagnosis has not yet been confirmed. Participants with one of the following two clinical presentations will be included: participants with evidence of de novo metastatic lung cancer or participants with evidence of de novo metastatic gastrointestinal cancer.

Participants may have undergone different levels of diagnostic workup prior to enrollment. Participants who have not had tissue biopsy performed prior to enrollment will be classified as 'basic workup' and those who have had tissue biopsy performed prior to enrollment will be classified as 'extended workup'.

During the diagnosis period, eligible participants will undergo liquid biopsy (FoundationOne® Liquid CDx assay; as per label) on blood samples. Blood samples will be tested using the FoundationOne® Liquid CDx assay at a central laboratory. In parallel, participants will undergo the standard of care diagnostic pathway, including tissue biopsy and histology workup, if not already done before enrollment, and molecular workup according to ESMO guidelines or national guidelines for each tumor type included in this study.

Once a complete pathologic diagnosis has been made, the investigator (or multidisciplinary team) can complete an anti-cancer treatment recommendation assessment. Anti-cancer treatment recommendation should follow current practice and professional guidelines based on the results provided by either liquid biopsy (as per label) or tissue biopsy/standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Participants presenting with a clinical diagnosis of advanced cancer, falling into one of the following two clinical presentations:

  i) De novo metastatic lung cancer as evidenced by imaging demonstrating a lung nodule/mass and objective evidence of a metastatic process; OR, ii) De novo metastatic gastrointestinal cancer as evidenced by imaging demonstrating a metastatic process in the abdomen/pelvis
* Participants who are treatment naïve for the metastatic setting under study
* Ability to comply with the study protocol
* Participants must either:

  i) Have a tissue biopsy intended/planned to confirm malignant disease and histology; OR, ii) Have a tissue biopsy already performed but pathology has not yet been finalized.

If a tissue biopsy has already been performed prior to ICF signature, then the subtyping of primary tumor may have already been assessed (i.e., for lung cancer TTF1, p40, and napsin A IHC staining may have already been performed).

Exclusion Criteria:

* Participants deemed not fit for treatment with systemic therapy
* Participants deemed not fit for tissue biopsy
* Participants with hematological neoplasm
* Participants with primary malignant neoplasm of the brain
* Participants with any previous molecular testing (NGS or other methods) e.g., all immunohistochemistry staining recommended by ESMO aiming to define the treatment decision (i.e., for lung cancer ALK, EGFR, and PD-L1 IHC staining must not have already been performed). Participants in which tissue biopsy and primary histotyping have been performed can be included in the study.
* Prior treatment for metastatic cancer with the exception of participants who have already been diagnosed and treated for cancer, other than the cancer type under study, who have no evidence of relapse
* History of malignancy within 5 years prior to screening, with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Median Time to Diagnosis | From the date of first request for biopsy (tissue or blood) by a healthcare professional to the date of complete pathologic diagnosis (up to 12 weeks)

SECONDARY OUTCOMES:
Median Time to Treatment Recommendation | From the date of first request for biopsy (tissue or blood) by a healthcare professional to the date of investigator's anticancer treatment recommendation (up to 12 weeks)
Number of Molecular Testing Failures | Up to 12 weeks
  Molecular testing failure is defined as cases in which the results of liquid biopsy or tissue biopsy/standard of care cannot be delivered to the treating physician.
Percentage of Participants in Which Comprehensive Genomic Profiling (CGP) Led to a Molecularly Guided Treatment Option (MGTO) Recommendation | Up to 12 weeks
  CGP refers to both the liquid biopsy and the standard of care diagnostic pathway.
Percentage of Participants Diagnosed with an Actionable Driver Mutation Who Did Not Receive a MGTO Because Anticancer Treatment Needed to Begin Before the CGP Results Were Available | Up to 12 weeks
Percentage of Participants With Concordant CGP Results Between the Liquid Biopsy and the Standard of Care Diagnostic Pathway on the Gene Alteration Level | Up to 12 weeks
Percentage of Participants in Which Treatment Recommendation Based on Molecular Data from the Liquid Biopsy Were the Same as That Based on the Standard of Care Diagnostic Pathway | Up to 12 weeks
Percentage of Participants in Which the MGTO Recommendation Issued Was Discordant Between the Liquid Biopsy Results and the Standard of Care Diagnostic Pathway Results | Up to 12 weeks
Incidence and Severity of Liquid Biopsy Sample Collection-Related Adverse Events | Up to 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- France (6):
  - Institut Sainte Catherine, Avignon
  - Hopital Marie Lannelongue, Le Plessis-Robinson
  - Centre Oscar Lambret, Lille
  - Centre Eugène Marquis, Rennes
  - CHU Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Gustave Roussy, Villejuif
- Germany (6):
  - Universitätsklinikum Hamburg-Eppendorf Onkologisches Zentrum Medizinische Klinik II, Hamburg
  - Med. Hochschule Hannover, Hanover
  - Universität Mannheim, Mannheim
  - Klinikum der LMU München, Campus Großhadern, Krebszentrum München, München
  - Asklepios Klinik Gauting, München-Gauting
  - Klinikum Stuttgart - Katharinenhospital, Stuttgart
- Italy (3):
  - Università degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Azienda Ospedaliero-Universitaria Dipartimento Interaziendale Di Oncologia, Udine, Friuli Venezia Giulia
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona, Veneto
- Spain (3):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Clinica Universidad de Navarra Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No